CLINICAL TRIAL: NCT01788488
Title: Impact of Measuring Serum Procalcitonin Levels on Duration of Antimicrobial Therapy in Critical Care Patients With Suspected Pneumonia
Brief Title: Procalcitonin Use in Pneumonia Patients in the Critical Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kent H. Gierhart, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-008835
Record Dates: First submitted 2013-01-25; First posted 2013-02-11 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Pneumonia
Keywords: procalcitonin; antimicrobial stewardship; pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Therapy (No Intervention)
- Procalcitonin-guided therapy (Experimental): Procalcitonin levels will be measured to determine when it is appropriate to discontinue antibiotic therapy.
  Interventions: Other: Use of procalcitonin as biomarker to guide therapy

INTERVENTIONS:
Other: Use of procalcitonin as biomarker to guide therapy
  Arms: Procalcitonin-guided therapy

SUMMARY:
The goal of the study is to determine the impact of procalcitonin (PCT)-guided therapy on duration of antibiotic therapy in critical care unit (CCU) patients with suspected pneumonia at Mayo Clinic Health System Eau Claire.

ELIGIBILITY:
Inclusion criteria:

* 18 years old
* admitted to critical care unit
* placed on pneumonia protocol

Exclusion criteria:

* patients who received outpatient antibiotic therapy within previous 21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Length of antibiotic therapy | Indefinite
  Participants will be followed for the entire time they are on antibiotics to treat pneumonia, an expected average of 30 total antibiotic days.

SECONDARY OUTCOMES:
Length of stay in critical care unit | Indefinite
  Participants will be followed for their entire length of stay in the critical care unit, an expected average of 7 days.
Cost | Once
  The average cost of antibiotics per patient, measured in US dollars, based on total antibiotic days.
Length of stay in the hospital | Indefinite
  Participants will be followed their entire length of stay in the hospital, an expected average of 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Gierhart, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System Eau Claire, Eau Claire, Wisconsin, United States

REFERENCES:
- [Background] Stolz D, Smyrnios N, Eggimann P, Pargger H, Thakkar N, Siegemund M, Marsch S, Azzola A, Rakic J, Mueller B, Tamm M. Procalcitonin for reduced antibiotic exposure in ventilator-associated pneumonia: a randomised study. Eur Respir J. 2009 Dec;34(6):1364-75. doi: 10.1183/09031936.00053209. Epub 2009 Sep 24. PMID 19797133
- [Background] Rice LB. The Maxwell Finland Lecture: for the duration-rational antibiotic administration in an era of antimicrobial resistance and clostridium difficile. Clin Infect Dis. 2008 Feb 15;46(4):491-6. doi: 10.1086/526535. PMID 18194098
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Christ-Crain M, Stolz D, Bingisser R, Muller C, Miedinger D, Huber PR, Zimmerli W, Harbarth S, Tamm M, Muller B. Procalcitonin guidance of antibiotic therapy in community-acquired pneumonia: a randomized trial. Am J Respir Crit Care Med. 2006 Jul 1;174(1):84-93. doi: 10.1164/rccm.200512-1922OC. Epub 2006 Apr 7. PMID 16603606
- [Background] Heyland DK, Johnson AP, Reynolds SC, Muscedere J. Procalcitonin for reduced antibiotic exposure in the critical care setting: a systematic review and an economic evaluation. Crit Care Med. 2011 Jul;39(7):1792-9. doi: 10.1097/CCM.0b013e31821201a5. PMID 21358400
- [Background] Agarwal R, Schwartz DN. Procalcitonin to guide duration of antimicrobial therapy in intensive care units: a systematic review. Clin Infect Dis. 2011 Aug;53(4):379-87. doi: 10.1093/cid/cir408. PMID 21810753
- [Background] Schuetz P, Albrich W, Mueller B. Procalcitonin for diagnosis of infection and guide to antibiotic decisions: past, present and future. BMC Med. 2011 Sep 22;9:107. doi: 10.1186/1741-7015-9-107. PMID 21936959
- [Background] Schuetz P, Chiappa V, Briel M, Greenwald JL. Procalcitonin algorithms for antibiotic therapy decisions: a systematic review of randomized controlled trials and recommendations for clinical algorithms. Arch Intern Med. 2011 Aug 8;171(15):1322-31. doi: 10.1001/archinternmed.2011.318. PMID 21824946
- [Background] Hayashi Y, Paterson DL. Strategies for reduction in duration of antibiotic use in hospitalized patients. Clin Infect Dis. 2011 May;52(10):1232-40. doi: 10.1093/cid/cir063. PMID 21507920
- [Background] Kook JL, Chao SR, Le J, Robinson PA. Impact of the use of procalcitonin assay in hospitalized adult patients with pneumonia at a community acute care hospital. Infect Control Hosp Epidemiol. 2012 Apr;33(4):424-6. doi: 10.1086/664764. PMID 22418643
- [Background] Kopterides P, Siempos II, Tsangaris I, Tsantes A, Armaganidis A. Procalcitonin-guided algorithms of antibiotic therapy in the intensive care unit: a systematic review and meta-analysis of randomized controlled trials. Crit Care Med. 2010 Nov;38(11):2229-41. doi: 10.1097/CCM.0b013e3181f17bf9. PMID 20729729
- [Background] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Background] Bouadma L, Luyt CE, Tubach F, Cracco C, Alvarez A, Schwebel C, Schortgen F, Lasocki S, Veber B, Dehoux M, Bernard M, Pasquet B, Regnier B, Brun-Buisson C, Chastre J, Wolff M; PRORATA trial group. Use of procalcitonin to reduce patients' exposure to antibiotics in intensive care units (PRORATA trial): a multicentre randomised controlled trial. Lancet. 2010 Feb 6;375(9713):463-74. doi: 10.1016/S0140-6736(09)61879-1. Epub 2010 Jan 25. PMID 20097417
- [Background] Li H, Luo YF, Blackwell TS, Xie CM. Meta-analysis and systematic review of procalcitonin-guided therapy in respiratory tract infections. Antimicrob Agents Chemother. 2011 Dec;55(12):5900-6. doi: 10.1128/AAC.00335-11. Epub 2011 Sep 26. PMID 21947386